CLINICAL TRIAL: NCT04478786
Title: What Are Ambulance Crews' Experiences of Using a Mechanical Chest Compression Device for Out-of-hospital Resuscitation? A Constructivist Qualitative Study Utilising Online Focus Groups
Brief Title: Ambulance Crews' Experiences of Using a Mechanical Chest Compression Device.
Status: Completed | Type: Observational
Sponsor: Northumbria University (Other)
Collaborators: Jolife AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 18018/275607
Record Dates: First submitted 2020-07-07; First posted 2020-07-21 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2020-07

CONDITIONS: Resuscitation
Keywords: Cardiopulmonary Resuscitation,; Resuscitation; Out of Hospital; Ambulance Crew; Mechanical Chest Compression Device; Qualitative; Experiences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Groups 1-4: An anticipated 3-8 participants who meet the inclusion criteria of being aged 18 or over, a employee of the local ambulance service, are employed as an operational ambulance crew member, irrespective of title and to have had experienced an out of hospital resuscitation where MCCD was used, irrespective of the type of device or their level of involvement, and who also volunteer and agree to take part in the online focus group.
  Interventions: Other: Focus group discussion

INTERVENTIONS:
Other: Focus group discussion — There is no intervention. This is a qualitative piece of work only.

SUMMARY:
Should a person have a cardiac arrest (where their heart stops beating) they require treatment of cardiopulmonary resuscitation (CPR). This includes providing chest compressions. Traditionally these compressions are provided by hand but mechanical chest compression devices (MCCD) have been investigated for use in out of hospital resuscitation attempts.

Research trials recruiting human participants have concluded recently. They all found no difference in survival outcomes when MCCD and manual compressions were compared.

Despite this, the latest expert review on MCCD suggests that MCCD can be a reasonable alternative to high quality manual compressions when these cannot be provided. MCCD continue to be used by Specialists in the local ambulance service and historically by those recruiting patients to a national multi centre trial of MCCD. There is another, as yet under-investigated element, and that is of ambulance crews' experiences of using such devices. Therefore it is a reasonable topic to investigate.

DETAILED DESCRIPTION:
This study will invite local United Kingdom (UK) National Health Service (NHS) operational ambulance crews to participate in a 1-2 hour online focus group discussion (a collective group discussion) about their experiences of using MCCD. The participants will be any operational ambulance crew member, employed by the local ambulance Trust and who had experience of using any type of MCCD. The focus groups will be audio recorded; participants will be aware of this when they choose to participate.

The aim of this research is to collect and report ambulance crews' experiences of using mechanical chest compression devices for out of hospital resuscitation attempts.

Ultimately there may of course be benefits for patients by exploring whether MCCD play a part in out of hospital resuscitations. Funding has been offered by a manufacturer one of the types of MCCD; they have had no involvement in the design or analysis of the study.

Once transcribed, the data will be analysed manually. The content of each focus group will be coded and then each participants' individual responses will be coded, first using open coding, then focused coding to identify emergent themes, before concluding with the categories that have been identified. The constant comparison method of data analysis will be used.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or over
* an employee of the local ambulance service
* employed as an operational ambulance crew member, irrespective of title
* to have experienced an out of hospital resuscitation where MCCD was used, irrespective of the type of device or their level of involvement.

Exclusion Criteria:

* not an employee of the local ambulance service
* have no experience of using a mechanical chest compression device at an out of hospital resuscitation
* the participant is unwilling to provide consent to participate
* the participant is unwilling to provide consent to be audio recorded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Operational ambulance crew employees of the local ambulance service
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2020-09-19 (Actual); Study Completion 2020-09-19 (Actual)

PRIMARY OUTCOMES:
Collect and report ambulance crews' experiences of using MCCDs for out-of-hospital resuscitation attempts. | 2 hours
  The transcribed discussions will be coded and then themes emerging from the data identified and developed. To do this I will use a constant comparison method of analysis. The presence or lack of consensus and reinforcement on certain topics will also be observed for.

OTHER OUTCOMES:
Does the use of MCCDs have any effect on, or facilitate, the team leader role at an out-of-hospital resuscitation attempt | 2 hours
  The transcribed discussions will be coded and then themes emerging from the data identified and developed. To do this I will use a constant comparison method of analysis. The presence or lack of consensus and reinforcement on certain topics will also be observed for.
Does providing mechanical versus manual chest compressions have an effect on how ambulance crews feel physically and emotionally after an out-of-hospital resuscitation attempt. | 2 hours
  The transcribed discussions will be coded and then themes emerging from the data identified and developed. To do this I will use a constant comparison method of analysis. The presence or lack of consensus and reinforcement on certain topics will also be observed for.

CONTACTS AND LOCATIONS:
Overall Officials: Richelle Duffy, PhD, Principal Investigator — Northumbria University
Locations (1):
- North East Ambulance Service NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Blair L, Duffy R. What are ambulance crews' experiences of using a mechanical chest compression device for out-of-hospital resuscitation? A constructivist qualitative study utilising online focus groups. Br Paramed J. 2022 Sep 1;7(2):24-30. doi: 10.29045/14784726.2022.09.7.2.24. PMID 36451709